CLINICAL TRIAL: NCT02424019
Title: A Phase 4 Safety Study of IOP Signals in Patients Treated With ILUVIEN® (Fluocinolone Acetonide Intravitreal Implant) 0.19 mg
Brief Title: Phase 4 IOP Signals Associated With ILUVIEN®
Acronym: PALADIN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alimera Sciences (Industry)
Responsible Party: Sponsor
Organization: ANI Pharmaceuticals (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M-01-15-004
Record Dates: First submitted 2015-04-18; First posted 2015-04-22 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Diabetic Macular Edema (DME)
MeSH Terms: interventions — Fluocinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ILUVIEN 0.19 MG (Experimental): All patients will receive ILUVIEN (Fluocinolone Acetonide Intravitreal Insert) 0.19 mg.
  Interventions: Drug: ILUVIEN 0.19 MG

INTERVENTIONS:
Drug: ILUVIEN 0.19 MG
  Other Names: Fluocinolone Acetonide Intravitreal Implant 0.19 mg

SUMMARY:
This study will assess the safety in patients treated with ILUVIEN, with primary focus on IOP.

DETAILED DESCRIPTION:
The specific objectives include the study of intraocular pressure (IOP) related data in patients who received ILUVIEN and how it relates to the patient's experiences following prior treatment with a course of corticosteroid which did not result in a clinically significant IOP elevation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible for treatment with ILUVIEN based on the Prescribing Information.

Exclusion Criteria:

* Patients who are unable to understand and sign the Informed Consent Form.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2015-05-06 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Intraocular Pressure | 36 months
  Intraocular pressure of the ILUVIEN treated eye

CONTACTS AND LOCATIONS:
Locations (41):
- United States (41):
  - Retina Consultants of Arizona, Phoenix, Arizona
  - Retina Centers, P.C., Tucson, Arizona
  - Retina and Macula Institute, Glendale, California
  - Atlantis Eye Care, Huntington Beach, California
  - Northern California Retina Vitreous Medical Group, Inc., Mountain View, California
  - Orange County Retina Medical Group, Santa Ana, California
  - Eye Care Center of Northern Colorado, Longmont, Colorado
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - Southeast Retina Center, P.C., Augusta, Georgia
  - Retina Consultants of Hawaii, ‘Aiea, Hawaii
  - Chicagoland Eye and Retina Foundation, Chicago, Illinois
  - The University of Illinois at Chicago, Chicago, Illinois
  - University Retina and Macula Associates, Oak Forest, Illinois
  - Illinois Retina Associates, SC, Oak Park, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Sabates Eye Center Research Division, Leawood, Kansas
  - Paducah Retinal Center, Paducah, Kentucky
  - Eye Associates of Northeast Louisiana, West Monroe, Louisiana
  - University of Maryland Eye Associates, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Wayne State University, Detroit, Michigan
  - Lifelong Vision Foundation, Chesterfield, Missouri
  - Discover Vision Centers, Independence, Missouri
  - Eyesight Ophthalmic Services, PA, Portsmouth, New Hampshire
  - New Jersey Retina, New Brunswick, New Jersey
  - Retina Associates of New Jersey, Teaneck, New Jersey
  - Joseph R. Podhorzer, MD PLLC, Brooklyn, New York
  - Ophthalmic Consultants of Long Island, Lynbrook, New York
  - Macula Care, New York, New York
  - Island Retina, Shirley, New York
  - Tulsa Retina Consultants, Tulsa, Oklahoma
  - Laurel Eye Clinic, Brookville, Pennsylvania
  - Pennsylvania Retina Specialist, PC, Camp Hill, Pennsylvania
  - Southeastern Retina Associates, PC, Kingsport, Tennessee
  - Retina Research Center, Austin, Texas
  - Valley Retina Institute, PA, McAllen, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Hampton Roads Retina Center, Chesapeake, Virginia
  - Virginia Retina Center, Warrenton, Virginia
  - Cascade Eye and Skin, University Place, Washington

REFERENCES:
- [Derived] Mansour SE, Kiernan DF, Roth DB, Eichenbaum D, Holekamp NM, Kaba S, Werts E. Two-year interim safety results of the 0.2 microg/day fluocinolone acetonide intravitreal implant for the treatment of diabetic macular oedema: the observational PALADIN study. Br J Ophthalmol. 2021 Mar;105(3):414-419. doi: 10.1136/bjophthalmol-2020-315984. Epub 2020 May 27. PMID 32461262